CLINICAL TRIAL: NCT01088204
Title: A Multicenter Randomized Phase II Clinical Trial of Laparoscopy Assisted Versus Open Distal Gastrectomy With D2 Lymph Node Dissection for Advanced Gastric Cancer
Brief Title: Feasibility Study of Laparoscopy-assisted D2 Distal Gastrectomy to Treat Advanced Gastric Cancer
Acronym: COACT_1001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Woo Kim, Head of Department of Gastric Cancer Surgery, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-09-448
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open distal gastrectomy (Active Comparator): open distal gastrectomy with D2 lymph node dissection for patients with advanced gastric cancer
  Interventions: Procedure: open distal gastrectomy
- laparoscopy assisted distal gastrectomy (Experimental): laparoscopy assisted distal gastrectomy with D2 lymph node dissection for patients with advanced gastric cancer
  Interventions: Procedure: laparoscopy assisted distal gastrectomy

INTERVENTIONS:
Procedure: laparoscopy assisted distal gastrectomy — laparoscopy assisted distal gastrectomy with D2 lymph node dissection for patients with advanced gastric cancer
  Other Names: LADG
  Arms: laparoscopy assisted distal gastrectomy
Procedure: open distal gastrectomy — open distal gastrectomy with D2 lymph node dissection for patients with advanced gastric cancer
  Other Names: ODG
  Arms: open distal gastrectomy

SUMMARY:
The purpose of this study is to evaluate the oncological feasibility of laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for advanced gastric cancer.

DETAILED DESCRIPTION:
To test oncological feasibility, compliance of nodal dissection was selected as a primary end point. When there are more than two missing nodal station(no lymph nodes in dissected area), it is defined as a non-compliant nodal dissection. Other secondary outcomes will be supplementary to evaluate feasibility of D2 dissection.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven primary gastric adenocarcinoma
* T2 or T3 or T4a, N0 or N1 or N2 or N3a (AJCC 7th), which is assessed by computed tomography (CT) scan - mid 1/3 or low 1/3 location
* No evidence of other distant metastasis
* not stump carcinoma,(vi) aged 20-80 year old
* performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* no prior treatment of chemotherapy or radiation therapy against any other malignancies, and no prior treatment for gastric cancer including endoscopic mucosal resection
* adequate organ functions defined as indicated below:

  * WBC 3000/mm3, WBC 12 000/mm3
  * Hb 8.0 g/dl without any transfusion 2 weeks before enrollment
  * Plt 100 000/mm3
  * AST 100 IU/l
  * ALT 100 IU/l
  * T.Bil 2.0 mg/dl
  * written informed consent

Exclusion Criteria:

* active double cancer (synchronous double cancer and metachronous double cancer within five disease-free years), excluding carcinoma in situ (lesions equal to intraepithelial or intramucosal cancer)
* pregnant or breast-feeding women
* severe mental disorder
* systemic administration of corticosteroids
* unstable angina or myocardial infarction within 6 months of the trial
* unstable hypertension
* severe respiratory disease requiring continuous oxygen therapy
* previous upper abdominal surgery except laparoscopic cholecystectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
noncompliance rate | postoperative 1 week
  A Case will be designated as "noncompliant" when there are more than one missing lymph node station according to the guidelines of "The Japanese Research Society for Gastric Cancer" (JRSGC) lymph node grouping

SECONDARY OUTCOMES:
Postoperative surgical complications | postoperative 1 day, 1 week, 1 months, 3 months, 6 months, 12 months
  Major and minor, and short term and long term complications related with surgery will be monitored and recorded according to classification of Accordion Severity Classification of Postoperative Complications; Expanded Classification.
operating time | operation day
  From skin incision to wound closure
time to first flatus | postoperative 1 week
  the day when a patient relieve gastrointestinal gas
number of retrieved lymph nodes | postoperative 1 week
number of retrieved lymph nodes at each stations | postoperative 1 week
proximal resection margin | postoperative 1 week
distal resection margin, | postoperative 1 week
unanimity rate of 3 randomly assigned laparoscopic gastric cancer surgeons | postoperative 3 months
  Three randomly assigned laparoscopic gastric cancer surgeons would evaluate the uneditted video and photoes and validate the lymph node dissection according to each stations.When the three surgeons agree that D2 lymph node dissection was performed, it is considered as unanimity.
3-year disease free survival | postoperative 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, MD,PhD, Principal Investigator — National Cancer Center, Korea
Locations (7):
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun, Chollanam Do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gyengsang National University Hospital, Jinju, Gyeongsangnam-do
  - Kyungpook national university hospital, Daegu
  - Dae Gu Veterans Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Kosin University Gospel Hospital, Pusan

REFERENCES:
- [Derived] Park YK, Yoon HM, Kim YW, Park JY, Ryu KW, Lee YJ, Jeong O, Yoon KY, Lee JH, Lee SE, Yu W, Jeong SH, Kim T, Kim S, Nam BH; COACT group. Laparoscopy-assisted versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: Results From a Randomized Phase II Multicenter Clinical Trial (COACT 1001). Ann Surg. 2018 Apr;267(4):638-645. doi: 10.1097/SLA.0000000000002168. PMID 28187041
- [Derived] Nam BH, Kim YW, Reim D, Eom BW, Yu WS, Park YK, Ryu KW, Lee YJ, Yoon HM, Lee JH, Jeong O, Jeong SH, Lee SE, Lee SH, Yoon KY, Seo KW, Chung HY, Kwon OK, Kim TB, Lee WK, Park SH, Sul JY, Yang DH, Lee JS. Laparoscopy Assisted versus Open Distal Gastrectomy with D2 Lymph Node Dissection for Advanced Gastric Cancer: Design and Rationale of a Phase II Randomized Controlled Multicenter Trial (COACT 1001). J Gastric Cancer. 2013 Sep;13(3):164-71. doi: 10.5230/jgc.2013.13.3.164. Epub 2013 Sep 30. PMID 24156036
- See also: National Cancer Center web site — http://ncc.re.kr